CLINICAL TRIAL: NCT05951517
Title: The Clinical Study of Mycophenolate Mofetil in Pediatric Refractory Gastrointestinal Henoch-Schonlein Purpura
Brief Title: Mycophenolate Mofetil in Gastrointestinal Henoch-Schonlein Purpura
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Weiping Tan, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-KY-021
Record Dates: First submitted 2023-06-19; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Henoch-Schönlein Purpura; Gastrointestinal Injury; Mycophenolate Mofetil
Keywords: Allergic purpura; complications,; renal involvement; gastrointestinal involvement; mycophenolate mofetil
MeSH Terms: conditions — IgA Vasculitis | interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mycophenolate mofetil in refractory gastrointestinal Henoch-Schönlein purpura (Experimental): patients who were resistant to steroid were treated with MMF
  Interventions: Drug: MMF

INTERVENTIONS:
Drug: MMF — MMF treat refractory gastrointestinal Henoch-Schönlein purpura
  Other Names: steroid

SUMMARY:
Henoch Schönlein purpura (HSP) is the most common type of vasculitis in children, with an incidence of ~10/100,000, whereas >90% of the patients develop symptoms at <10 years of age. Although HSP is generally a self-limiting disease, it may also lead to severe complications, such as intestinal intussusception, infarction and perforation, as well as end-stage renal disease. The management of HSP includes symptomatic treatment and immunosuppressive therapy in certain patients. Previous retrospective studies have reported that most patients with gastrointestinal (GI) symptoms may benefit from early usage of glucocorticoid, whereas there are still a part of HSP patients with GI did not achieved remission after administering of steroid. Therefore, the aim of the present study was to investigate the clinical features of refractory GI HSP and the clinical outcome of mycophenolate mofetil in these patients.

DETAILED DESCRIPTION:
the aim of the present study was to investigate the clinical features of refractory GI HSP and the clinical outcome of mycophenolate mofetil in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages range from 3 to 18 years old;
2. Patients who meet the diagnostic criteria for HSP and involve the digestive tract: acute diffuse abdominal colic, including intussusception and gastrointestinal bleeding, appears during the course of the disease or is found on physical examination;
3. Refractory gastrointestinal type HSP: treated with Intravenous corticosteroid 2 mg/kg/d for 3 days without effecacy or relapsed during the attenuation of corticosteroid
4. Parents or guardians agree to treatment and sign a written informed consent form.

Exclusion Criteria:

1. Patients who are allergic to MMF;
2. Patients with severe diseases: such as systemic malignancies, heart failure, liver and renal failure, Immune deficiency, severe infectious diseases, organ transplant surgery, or other current indications for emergency surgery;
3. Patients with other digestive system diseases;
4. Those who have previously used MMF clinical trials;
5. Other situations the researcher thought inappropriate to participate in the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Abdominal pain, hematemesis and bloody stools | 6 months
  assessed by checklist

SECONDARY OUTCOMES:
count of red blood cells in Stool | 6 months
  Test for every week

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Tan, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China